CLINICAL TRIAL: NCT06489691
Title: Comparative Study of 6-minute Walk Distance (6MWD) in Patients With High Altitude Pulmonary Hypertension Permanently Residing Above 2500 Meters When Assessed Near Resident High Altitude (HA) at 3200m vs. at Low Altitude (LA) 760m
Brief Title: High Altitude Residents With High Altitude Pulmonary Hypertension (HAPH), 6MWT Assessed at High Altitude (3200m) vs Low Altitude (760m)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: HAPH_HAvsLA_6MWT
Record Dates: First submitted 2024-06-28; First posted 2024-07-08 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: High Altitude Pulmonary Hypertension
Keywords: Pulmonary Hypertension; Hypoxia; High Altitude; 6-Minute Walk Test
MeSH Terms: conditions — Pulmonary edema of mountaineers; Hypertension, Pulmonary; Hypoxia; Altitude Sickness

STUDY DESIGN:
Intervention Model Description: Each highlander with HAPH will perform a 6 MWT at 3200 m and at 760 m according to a prospective study design
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Assessments at 3200 m and 760 m, respectively (Experimental): Participants will have a 6-minute walk distance (6MWD) assessment near their resident altitude at 3200 m and after relocation to 760 m after 1 and 7 days.
  Interventions: Other: 6-minute walk test (6MWT)

INTERVENTIONS:
Other: 6-minute walk test (6MWT) — 6-minute walk test (6MWT) will be performed according to clinical standards

SUMMARY:
To study the effect of relocation from 3200m (Aksay) to 760m (Bishkek) in highlanders with High Altitude Pulmonary Hypertension (HAPH) who permanently live >2500m on 6-minute walk distance (6MWD)

DETAILED DESCRIPTION:
This research in highlanders with HAPH diagnosed by echocardiography and defined by a RV/RA >30 mmHg who permanently live at HA >2500 m will perform a 6-minute walk distance test near their living altitude in Aksay at 3200 m and on day 2 and 7 at 760 m after relocation

ELIGIBILITY:
Inclusion Criteria:

* Permanently living >2500 m
* HAPH diagnosed with a minimum RV/RA of 30 mmHg assessed by echocardiography at an altitude of 3200 m
* Written informed consent

Exclusion Criteria:

* Highlanders who cannot follow the study investigations,
* Patients with moderate to severe concomitant lung disease (FEV1<70% or forced vital capacity <70%), severe parenchymal lung disease, heavy smoking >20 cigarettes/day or >20 pack-years.
* Coexistent unstable systemic hypertension or coronary artery disease that required adjustment of medication within the last 2 months
* Regular use of medication that affects control of breathing (benzodiazepines, opioids, acetazolamide)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2024-07-02 (Actual); Primary Completion 2024-09-27 (Actual); Study Completion 2024-09-27 (Actual)

PRIMARY OUTCOMES:
6-minute walk distance (6MWD) on day 2 of relocation to 760 m | day 2 at 760 m compared to 3200 m
  Change in 6MWD in meter between LA (760 m) vs HA (3200 m)

SECONDARY OUTCOMES:
6-minute walk distance (6MWD) on day 7 of relocation to 760 m | day 7 at 760 m compared to 3200 m
  6-minute walk distance (6MWD) in meter between LA (760 m) and HA (3200 m)
Arterial oxygen saturation by pulseoximetry (SpO2) at rest and at peak 6MWD on day 2 of relocation to 760 m | day 2 at 760 m compared to 3200 m
  Change in SpO2 in % between LA (760 m) vs HA (3200 m)
Arterial oxygen saturation by pulseoximetry (SpO2) at rest and at peak 6MWD on day 7 of relocation to 760 m | day 7 at 760 m compared to 3200 m
  Change in SpO2 in % between LA (760 m) vs HA (3200 m)
Heart rate at rest and at peak 6MWD on day 2 of relocation to 760 m | after the first night at LA (760 m)
  Change in hear rate in bpm between LA (760 m) vs HA (3200 m)
Heart rate at rest and at peak 6MWD on day 7 of relocation to 760 m | day 7 at 760 m compared to 3200 m
  Change in hear rate in bpm between LA (760 m) vs HA (3200 m)
Blood pressure at rest and at 6MWD on day 2 of relocation to 760 m | day 2 at 760 m compared to 3200 m
  Change in blood pressure in mmHg between LA (760 m) vs HA (3200 m)
Blood pressure at rest and at 6MWD on day 7 of relocation to 760 m | day 7 at 760 m compared to 3200 m
  Change in blood pressure in mmHg between LA (760 m) vs HA (3200 m)
Borg Dyspnea scale at end 6MWT on day 2 of relocation to 760 m | day 2 at 760 m compared to 3200 m
  Change of the Borg CR10 dyspnea scale at end of the 6MWT after the first night at LA (760 m) vs HA (3200 m)
Borg Dyspnea scale at end 6MWT on day 7 of relocation to 760 m | day 7 at 760 m compared to 3200 m
  Change of the Borg CR10 dyspnea scale at end of the 6MWT after seven nights at LA (760 m) vs HA (3200 m)
Borg leg fatigue scale at end 6MWT on day 2 of relocation to 760 m | day 2 at 760 m compared to 3200 m
  Change of the Borg CR10 leg fatigue scale at end of the 6MWT after the first night at LA (760 m) vs HA (3200 m)
Borg leg fatigue scale at end 6MWT on day 7 of relocation to 760 m | day 7 at 760 m compared to 3200 m
  Change of the Borg CR10 leg fatigue scale at end of the 6MWT after seven nights at LA (760 m) vs HA (3200 m)

CONTACTS AND LOCATIONS:
Overall Officials: Talant M Sooronbaev, Prof. Dr., Principal Investigator — National Center of Cardiology and Internal Medicine named after academician M.Mirrakhimov; Silvia Ulrich, Prof. Dr., Principal Investigator — University Hospital Zurich, Department of Pulmonology
Locations (1):
- Aksay Medical Center, Aksay Plateau, Naryn, Kyrgyzstan, Kyrgyzstan

IPD SHARING:
Plan to Share IPD: Undecided